CLINICAL TRIAL: NCT00402610
Title: A Randomized Trial of Three Regimens to Prevent Tuberculosis in HIV-Infected Patients With Anergy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sociedad Andaluza de Enfermedades Infecciosas (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GAEI 94/0071a; FIS 94/0071A
Record Dates: First submitted 2006-11-18; First posted 2006-11-22 (Estimated); Last update posted 2008-10-24 (Estimated); Status verified 2006-11

CONDITIONS: HIV Infections; Tuberculosis
Keywords: HIV; Tuberculosis; Chemoprophylaxis; Anergy; AIDS
MeSH Terms: conditions — HIV Infections; Tuberculosis; Acquired Immunodeficiency Syndrome | interventions — Isoniazid; Rifampin; Pyrazinamide

INTERVENTIONS:
Drug: isoniazid, rifampin + isoniazid, rifampin + pyrazinamide or not treatment

SUMMARY:
INTRODUCTION. To evaluate the efficacy of three regimens of prophylactic therapy for tuberculosis in HIV-infected patients with anergy. METHODS. Prospective, multi-center, randomized, comparative, and open clinical trial. Anergy was defined as absence of induration in response to three antigens (PPD, Candida albicans and parotiditis antigen) applied by the Mantoux method. Patients were randomized into one of the following prophylactic treatment groups: isoniazid for six months (6H), rifampin plus isoniazid for three months (3RH), rifampin plus pyrazinamide for two months (2RZ) or no treatment (NT). After completion of treatment, patients were followed up for two years.

DETAILED DESCRIPTION:
This study is a controlled, open, randomized, multi-center clinical trial. The study was authorized by the Clinical Research Ethics Committee of all participating centers and informed written consent was obtained from all the patients included. The cutaneous anergy was defined by the absence of a reaction (0 mm) to skin reactivity tests with tuberculin, Candida albicans, and parotiditis antigens 72 hours after inoculation. The patients were randomzed into one of the following four groups: isoniazid for 6 months (6H), rifampin plus isoniazid for 3 months (3RH), rifampin plus pyrazinamide for 2 months (2RZ) or no treatment (NT). All of the participating subjects underwent a basal study that included clinical and epidemiological history, chest x-ray, hemogram, analysis of serum creatinine concentrations, uric acid, AST, ALT, alkaline phosphatase, and total bilirubin, as well as a CD4+ T-lymphocyte count.During prophylactic treatment, patients were evaluated every 15 days for the first two months and monthly thereafter. At each check-up it was determined whether or not the patient was following the treatment properly and whether there were any adverse effects. Therapeutic completion was defined as taking at least 80% of the total prescribed dosages.Chemoprophylaxis was discontinued whenever a patient requested to do so or for any of the following reasons: appearance of Grade 3 or 4 side effects that could be attributed to the drugs used in the study; increases in AST and/or ALT values of three times or more their basal values; development of TB; or diagnosis of any disease that made interruption of the treatment advisable.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection confirmed by ELISA and Western blot
* Age between 18 and 65 years
* Life expectancy greater than two years
* Cutaneous anergy defined by the absence of a reaction (0 mm) to skin reactivity tests with tuberculin, Candida albicans, and parotiditis antigens 72 hours after inoculation.

Exclusion Criteria:

* Presence of active tuberculosis
* Background of previous antituberculosis therapy or chemoprophylaxis
* Presence of symptoms or signs suggesting pulmonary or extra-pulmonary tuberculosis
* History of hypersensitivity to the drugs used in the study (isoniazid, rifampin or pyrazinamide)
* Aspartate-aminotransferase and/or alanine-aminotransferase plasma concentrations more than or equal to four times their normal values, total bilirubin more than 2 mg/ml, and/or creatinine more than 2 mg/ml
* Pregnancy
* Undergoing treatment incompatible with any of the drugs used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332
Dates: Start 1994-01; Study Completion 1998-12

PRIMARY OUTCOMES:
Development of tuberculosis

SECONDARY OUTCOMES:
Suspension of chemoprophylaxis due to adverse effects
Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rivero, MD PhD, Study Chair — Hospital Universitario Reina Sofía, Córdoba, Spain; Luis Lopez-Crtés, MD, PhD, Principal Investigator — Hospital Universitario Virgen del Rocío, Sevilla, Spain; Rafael Castillo, MD, Principal Investigator — 3 Sección de Enfermedades Infecciosas. Hospital Clínico Universitario San Cecilio. Avda. Dr. Oloriz 16. 18012 Granada; José Verdejo, MD, Principal Investigator — Servicio de Enfermedades Infecciosas. Hospital Carlos III. Sinesio Delgado 10. 28029 Madrid; Miguel Angel García, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Carlos Haya. Avda. Carlos Haya s/n. 29010 Málaga.; Felipes Diez, MD, Principal Investigator — Servicio de Medicina Interna. Hospital Torrecárdenas. Paraje de Torrecárdenas s/n. 04009 Almería.; Jose Carlos Escribano, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Universitario Puerta del Mar. Avda. Ana de Viya, 21. 11009 Cádiz. Spain; Jesús Canueto, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Punta Europa de Algeciras. Ctra de Getares s/n. 11207 Algeciras (Cádiz)., Spain; Manuel Marquez, MD, Principal Investigator — Unidad de Enfermedades Infecciosas. Hospital Universitario Virgen de la Victoria, Campus Universitario Teatinos s/n. 29010 Málaga.; Juan Jose Hernandez, MD, Principal Investigator — Unidad de Enfermedades Infecciosas. Hospital Ciudad de Jaén, Avda del Ejército Español, 10. 23007 Jaén, Spain.; Juan Pasquau, MD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Universitario Virgen de las Nieves. Avda de las Fuerzas Armadas, 2. 18014 Granada, Spain.; Fernando Lozano, MD PhD, Principal Investigator — Sección de Enfermedades Infecciosas. Hospital Universitario Virgen de Valme. Ctra. de Cádiz s/n. 41012 Sevilla, Spain
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

REFERENCES:
- [Result] Rivero A, Lopez-Cortes L, Castillo R, Lozano F, Garcia MA, Diez F, Escribano JC, Canueto J, Pasquau J, Hernandez JJ, Polo R, Martinez-Marcos FJ, Kindelan JM, Rey R; Grupo Andaluz para el estudio de las Enfermedades Infecciosas (GAEI). [Randomized trial of three regimens to prevent tuberculosis in HIV-infected patients with anergy]. Enferm Infecc Microbiol Clin. 2003 Jun-Jul;21(6):287-92. doi: 10.1016/s0213-005x(03)72942-5. Spanish. PMID 12809582